CLINICAL TRIAL: NCT06759649
Title: A First-in-Human, Phase 1 Dose Escalation and Dose Expansion Trial to Assess the Safety and Tolerability of COM503 as Monotherapy and in Combination Therapy in Participants With Advanced Solid Malignancies
Brief Title: A Clinical Trial to Assess COM503 in Participants With Advanced Solid Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Compugen Ltd (Industry)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CPG-05-101
Record Dates: First submitted 2024-12-19; First posted 2025-01-06 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-09

CONDITIONS: Neoplasm; Cancer, Malignant Tumors
Keywords: first-in-human; oncology; monoclonal antibody; immunotherapy
MeSH Terms: conditions — Neoplasms | interventions — zimberelimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1, A-1 (Experimental): Monotherapy Dose Escalation
  Interventions: Drug: COM503
- Part 1, A-2 (Experimental): Backfill
  Interventions: Drug: COM503
- Part 1, B (Experimental): Dose escalation, COM503 in combination with a fixed dose of zimberelimab.
  Interventions: Drug: COM503; Drug: Zimberelimab
- Part 2, A (Experimental): Dose expansion, COM503 monotherapy
  Interventions: Drug: COM503
- Part 2, B (Experimental): Dose expansion, COM503 in combination with a fixed dose of zimberelimab.
  Interventions: Drug: COM503; Drug: Zimberelimab

INTERVENTIONS:
Drug: COM503 — Intravenous Infusion
Drug: Zimberelimab — Intravenous infusion
  Arms: Part 1, B; Part 2, B

SUMMARY:
The overall goal of this first-in-human (FIH) clinical trial is to learn about the safety and dosing of COM503 when given alone or in combination with zimberelimab in participants with advanced solid tumors.

The primary objectives of this study are:

* To assess the safety and tolerability of COM503 as monotherapy and COM503 in combination with zimberelimab in participants with advanced solid tumors.
* To identify the maximum tolerated dose (MTD) / maximum administered dose (MAD) and/or the recommended phase 2 dose (RP2D) of COM503 as monotherapy and in combination with zimberelimab in participants with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Participants with histologically/cytologically confirmed advanced recurrent or metastatic solid tumor malignancy
* Part 1 (dose escalation): Participants must have had disease progression on or following all available standard of care (SOC) therapies known to confer clinical benefit.
* Part 2 (dose expansion): Participants may be enrolled following disease progression that has progressed after at least 1 available standard therapy; or for whom standard therapy has proven to be ineffective or intolerable or is considered inappropriate; or for whom a clinical trial of an investigational agent is a recognized SOC.
* Participants must have a solid tumor measurable by computed tomography (CT) or magnetic resonance imaging (MRI) as per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) criteria by investigator assessment

Exclusion Criteria:

* History of another malignancy within 2 years prior to the first trial intervention administration (unless the malignancy was treated with curative intent with low risk of recurrence [e.g., nonmelanoma skin cancer, histologically confirmed complete excision of carcinoma in situ, or similar] which are allowed to enroll).
* Therapy with Immunosuppressive doses of systemic medications, such as steroids (doses >10 mg/day prednisone or equivalent daily) within 2 weeks before trial intervention administration
* Have known active central nervous system (CNS) metastases and/or leptomeningeal disease (LMD).
* Active and clinically relevant bacterial, fungal, or viral infection that is not controlled or requires systemic antibiotics, antifungals, or antivirals, respectively.
* Ascites or pleural effusion that is symptomatic and/or requiring drainage within 2 weeks prior to the first trial intervention administration.
* Have active hepatitis B virus (HBV) or hepatitis C virus (HCV), or participants with human immunodeficiency virus (HIV).
* Any medical condition that, in the investigator's or sponsor's opinion, poses an undue risk to the participant's participation in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2027-11-22 (Estimated); Study Completion 2027-11-22 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety profile of COM503 as monotherapy in participants with advanced malignancies. | from the first dose of COM503 to the earlier of 90 days following the last dose of COM503 and/or zimberelimab or start of a new anticancer therapy.
  Number of participants in monotherapy cohorts with treatment-related adverse events as assessed by CTCAE v4.0
To evaluate the safety profile of COM503 as monotherapy in participants with advanced malignancies. | from the first dose of COM503 to the earlier of 90 days following the last dose of COM503 and/or zimberelimab or start of a new anticancer therapy.
  Number of participants in monotherapy cohorts with treatment-related serious adverse events as assessed by CTCAE v4.0
To evaluate the safety profile of COM503 in combination with zimberelimab in participants with advanced malignancies | from the first dose of COM503 in combination with zimberelimab to the earlier of 90 days following the last dose of COM503 and/or zimberelimab or start of a new anticancer therapy.
  Number of participants in combination cohorts with treatment-related adverse events as assessed by CTCAE v4.
To evaluate the safety profile of COM503 in combination with zimberelimab in participants with advanced malignancies | from the first dose of COM503 to the earlier of 90 days following the last dose of COM503 and/or zimberelimab or start of a new anticancer therapy.
  Number of participants in combination cohorts with treatment-related serious adverse events as assessed by CTCAE v4.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (7):
  - Yale- New Haven Hospital- Yale Cancer Center, New Haven, Connecticut
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - START Midwest, Grand Rapids, Michigan
  - The West Clinic, PLCC dba West Cancer Center, Germantown, Tennessee
  - NEXT Oncology San Antonio, San Antonio, Texas
  - START, San Antonio, Texas
  - NEXT Oncology Virginia, Fairfax, Virginia
- Rambam Health Care Campus, Haifa, Israel, Israel

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol